CLINICAL TRIAL: NCT00100152
Title: A Phase I Study of a Gamma Secretase Inhibitor for Adult and Pediatric Patients With Relapsed or Refractory Acute T-Cell Lymphoblastic Leukemia and Lymphoma
Brief Title: A Notch Signalling Pathway Inhibitor for Patients With T-cell Acute Lymphoblastic Leukemia/Lymphoma (ALL)(0752-013)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0752-013; 2004_097
Record Dates: First submitted 2004-12-23; First posted 2004-12-24 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Leukemia, Lymphoblastic, Acute, T-cell; Myelogenous Leukemia; Chronic Lymphocytic Leukemia; Myelodysplastic Syndromes
Keywords: Relapsed or refractory T-cell ALL acute lymphoblastic/leukemia; Relapsed/refractory T-cell acute Lymphoblastic/leukemia; Acute/chronic myelogenous leukemia; Poor-risk myelodysplasia
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid; Leukemia, Lymphocytic, Chronic, B-Cell; Myelodysplastic Syndromes; Recurrence; Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — 3-(4-((4-chlorophenyl)sulfonyl)-4-(2,5-difluorophenyl)cyclohexyl)propanoic acid

INTERVENTIONS:
Drug: MK0752, (Notch Inhibitor)

SUMMARY:
A Notch signalling pathway inhibitor study in pediatric and adult patients with relapsed (worsening) or refractory (not responding to treatment) T-cell acute lymphoblastic leukemia/lymphoma (T-ALL).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically documented precursor T-cell acute lymphoblastic leukemia/lymphoma (T-ALL), relapsed or refractory to standard therapy, or not be a candidate for standard myelosuppressive chemotherapy due to age or comorbid disease.
* Patient must have performance status <2 on the ECOG performance status for patients >16 years old; Lansky performance level >50 for patients 12 months to less than or equal to 16 years old.
* Patient must have adequate renal and liver function as indicated by the laboratory values performed within 14 days of receiving the first dose of study drug.
* Patient must have fully recovered from any chemotherapy and be greater than 2 weeks from radiotherapy, immunotherapy, or systemic steroid therapy with the exception of hydroxyurea, intrathecal therapy, or immunosuppressant therapy for chronic graft-versus-host disease prophylaxis following allogeneic bone marrow transplant.
* Patient must be greater than 2 months following bone marrow or peripheral blood stem cell transplantation and off all immunosuppressant therapy (with the exception of patients taking immunosuppressant therapy for chronic graft-versus-host disease prophylaxis following allogeneic bone marrow transplant).
* Men and women of reproductive potential must use an effective contraceptive method while enrolled in the study.
* Patient or the patient's legal representative must be able to understand the study and give written informed consent.

Exclusion Criteria:

* Patient has had treatment with any investigational therapy during the preceding 30 days.
* Patient has uncontrolled congestive heart failure, angina, or had a myocardial infarction in the preceding 3 months.
* Patient has known hypersensitivity to the components of study drug, its analogs, or to allopurinol.
* Patient has active or uncontrolled infection.
* Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Patient is pregnant or lactating.
* Patient has any other severe concurrent disease which would make the patient inappropriate for entry into this study.
* Patient is known to be HIV positive or who has an AIDS-related illness.
* Patients with a "currently active" second malignancy, other than non-melanoma skin cancer should not be enrolled.
* Patient has isolated CNS disease.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2005-02; Primary Completion 2006-09 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC